CLINICAL TRIAL: NCT06961344
Title: An Open-label Extension Study Evaluating the Safety of Zagociguat in Participants With MELAS Who Completed TIS6463-203
Brief Title: An Open-label Extension Safety Study of MELAS Patients Who Completed TIS6463-203 (PRIZM)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS6463-204
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mitochondrial Encephalopathy, Lactic Acidosis and Stroke-Like Episodes (MELAS Syndrome)
Keywords: MELAS
MeSH Terms: conditions — Mitochondrial encephalopathy; Acidosis, Lactic; MELAS Syndrome

STUDY DESIGN:
Intervention Model Description: An open-label, single-group assignment extension study.
  Eligible patients will be entered into a single treatment sequence. The treatment period will last for the shortest of the following: 104 weeks; regulatory approval and commercial availability of zagociguat in the participant's respective country; or termination of the clinical development of zagociguat in MELAS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zagociguat 15mg (Experimental): Participants receive zagociguat 15 mg once a day (QD) for the duration of the study.
  Interventions: Drug: zagociguat 15mg

INTERVENTIONS:
Drug: zagociguat 15mg — once daily oral tablets
  Other Names: IW-6463; CY6463

SUMMARY:
The goal of this clinical trial is to evaluate the long-term safety and tolerability of zagociguat in patients with MELAS who completed study medication treatment in the lead-in study TIS6463-203. TIS6463-204 is evaluating zagociguat in an open-label extension study at the daily dose of 15mg. The study medication is a once daily oral table and will be provided at the clinic and/or shipped to the participant's home. Study assessments will be conducted during clinic visits which will occur at three months and then at six months. Thereafter, clinic visits will occur every six months.

DETAILED DESCRIPTION:
On Screening Visit Day -1 (which corresponds to Period 2 Week 12 Visit from lead-in study TIS6463-203), participants will sign the informed consent form, be confirmed eligible for this open-label extension study and undergo Screening Visit assessments. Eligible participants will begin dosing the next day on Day 1 (there is no Day 0) at home. Participants will have a 3-month visit and 6-month study visit at the clinic and thereafter will have a clinic visit every 6 months. Participants should have a Follow-up Visit 4 (+1) weeks after zagociguat discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form (ICF).
2. Completed TIS6463-203 treatment through the Period 2 Week 12 Visit.
3. Agrees to follow lifestyle restrictions.
4. Other criteria per the protocol.

Exclusion Criteria:

1. Any medical condition or clinical finding that, per investigator judgement, would preclude safe study participation and/or completion of all trial requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) | Day 1 through the Follow-up for treatment period 4 weeks after last dose of study medication.
  TEAEs are any untoward event that may or may not be related to study medication.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - UC San Diego - Altman Clinical and Translational Research Institute, La Jolla, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Rare Disease Research, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai - Ichan School of Medicine, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - UT Health Houston, Houston, Texas
- Royal Melbourne Hospital, Melbourne, Victoria, Australia
- LMU Klinikum, Friedrich-Baur-Institute, Department of Neurology, Munich, Germany
- Neurologic Institute Carlo Besta of Milan, Milan, Italy
- United Kingdom (2):
  - University College London Hospital. The National Hospital for Neurology and Neurosurgery, Centre for Neuromuscular Diseases, London
  - The Newcastle upon Tyne NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No